CLINICAL TRIAL: NCT00693355
Title: Effects of Butyrate Enemas on Colonic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Fred Troost, University of Maastricht
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MEC 05-137
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: gut health
MeSH Terms: interventions — Butyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): sodium butyrate
  Interventions: Other: Sodium butyrate
- 2 (Placebo Comparator): NaCl
  Interventions: Other: NaCl

INTERVENTIONS:
Other: Sodium butyrate — sodium butyrate
  Arms: 1
Other: NaCl — NaCl
  Arms: 2

SUMMARY:
Short chain fatty acids (mainly acetate, propionate and butyrate) are produced in the large intestine by bacterial fermentation of unabsorbed carbohydrates, such as dietary fibers. Mainly butyrate is an important energy source of the mucosa and has a pivotal role in the regulation of mucosal proliferation, immune function and mucosal protection.

High fiber diets increase the concentrations of colonic butyrate, what has often been proposed as one of its protective mechanisms. Furthermore, butyrate enemas have been proved effective in the treatment of ulcerative colitis. In the present study the direct effects of butyrate on the distal colon will be studied in 30 healthy volunteers using rectal enemas. The study has been divided into two parts, each part studying different parameters, which interfere when measured synchronously and, therefore, need to be studied separately.

A. The effects of butyrate enemas on colonic permeability (n=15) B. The effects of butyrate enemas on parameters of colonic defense, integrity and inflammation (n=15) The effects of butyrate will be studied in a healthy and in a stressed colon. This way the protective effects of butyrate on intestinal stress can be studied. Prior to the main study, two small pilot studies will be carried out. In the first pilot study the retrograde spread of a rectal enema will investigated (n=2). In the second pilot study the dose and the type of a suitable stressor that will induce reversible damage to intestinal mucosa will be determined (n=12).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old
* Good medical health according to a standard medical questionnaire
* Regular defecation pattern (at least once daily)

Exclusion Criteria:

* Use of medication other than oral anticonceptives
* Calcium supplementation (during the study)
* Caloric restriction diet (during the study)
* Excessive drinking (>2 alcoholic consumptions a day)
* Drug abuse in the past six months and during the study
* Infectious disease (1 month prior to the study)
* Pregnant or lactating women
* Problems with urinary tract
* History of gastrointestinal complaints or disease(s)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
inflammatory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Fred Troost, PhD, Principal Investigator — Maastricht University
Locations (1):
- University of Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Hamer HM, Jonkers DM, Bast A, Vanhoutvin SA, Fischer MA, Kodde A, Troost FJ, Venema K, Brummer RJ. Butyrate modulates oxidative stress in the colonic mucosa of healthy humans. Clin Nutr. 2009 Feb;28(1):88-93. doi: 10.1016/j.clnu.2008.11.002. Epub 2008 Dec 23. PMID 19108937